CLINICAL TRIAL: NCT06878690
Title: Characterization of Sleep Disorders in Patients With Specific Learning Disabilities According to Age, Sex, Associated Comorbidities and Treatments
Brief Title: Sleep Disorders in Specific Learning Disabilities
Acronym: DYSOM
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0276; 2024-A01674-43 (Other: ID-RCB)
Record Dates: First submitted 2025-03-05; First posted 2025-03-17 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Specific Learning Disability; Sleep; Sleep Disorder (Disorder); ADHD
Keywords: Specific learning disabilities; Sleep; ADHD; Paediatric
MeSH Terms: conditions — Sleep Wake Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children: Children (4 < 18 years old) with specific learning disabilities, associated or not with others medical condition
  Interventions: Other: Online Questionnaire
- Adult: Adult (> 18 years old) with specific learning disabilities, associated or not with others medical condition
  Interventions: Other: Online Questionnaire

INTERVENTIONS:
Other: Online Questionnaire — Completion of an online questionnaire via the secure RedCap platform

SUMMARY:
Specific learning disorders, or SLD, are cognitive and behavioral conditions that emerge during childhood and involve significant difficulties in acquiring and performing specific intellectual, motor, language, and social functions. These disorders impact personal, social, academic, and professional functioning throughout life. In France, between 6% and 8% of the population, including both children and adults, are affected by at least one type of SLD.

SLD are also frequently associated with Attention Deficit Hyperactivity Disorder (ADHD), with prevalence rates ranging from 33% to 70%, depending on the study. This comorbidity leads to more severe attention and learning difficulties than when ADHD or SLD occur independently.

ADHD is a common neurodevelopmental disorder that affects cognitive attentional processes, with or without hyperactivity. It is estimated to affect approximately 5.3% of children and adolescents worldwide and about 3% of adults.

The assessment of these disorders is conducted through a neuropsychological evaluation, which determines the type and severity of cognitive impairments.

Several studies report that 55% to 74% of children with ADHD experience sleep difficulties.

To date, only two studies have examined the prevalence of sleep disorders among children with SLD disorders. One of these studies focused exclusively on dyslexia, with or without ADHD. The results revealed significantly higher scores among dyslexic children compared to controls when completing sleep disorder assessment questionnaires (SDSC). The main difficulties were related to "sleep onset and maintenance disorders," "sleep-related breathing disorders," and "wakefulness disorders." The second study, using the same questionnaire, compared children with ADHD, SLD disorders, and both combined. The group with co-existing SLD and ADHD disorders exhibited significantly more sleep disturbances than the other groups, primarily sleep onset and maintenance disorders.

Despite the importance of these studies, they focused only on sleep disorders associated with dyslexia, without considering other learning disorders such as dyspraxia, dyscalculia, or dysgraphia. Furthermore, when ADHD was taken into account, the studies did not differentiate between its various forms, limiting the interpretation of the results. Additionally, no research has tracked the evolution of sleep disorders in the SLD +/- ADHD population from childhood through adolescence and into adulthood.

In this study, the investigators aim to evaluate sleep disorders in the SLD population (with or without ADHD) in France through online questionnaires. These questionnaires will be offered to 1,000 children (aged ≥4 years) and adults diagnosed with at least one specific learning disorder.

Primary Objective:

The main objective of this study is to assess the frequency and nature of sleep disorders in patients (both adults and children) with specific learning disorders, with or without ADHD.

Secondary Objectives:

* Characterize the "SLD" patient population in France by considering age and gender:

  o Determine the prevalence of co-morbidities, such as: ADHD Anxiety and depressive disorders Other reported medical conditions
  * Assess the types of care provided (medication or other) for both children and adults
  * Determine the frequency of SLD in a familial context
* Identify whether the following factors are associated with a higher frequency of sleep disorders:

  * Single SLD vs. multiple SLD
  * The presence of ADHD, anxiety-depressive disorders, or other medical conditions alongside SLD
  * Demographic characteristics (age, gender, etc.)
  * Family history of SLD among relatives (parents and siblings)
  * Medication use

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents and adults with a specific learning disability (dyslexia, dysorthography, dyscalculia, dysgraphia, dyspraxia, dysphasia).
* ≥ 4 ans

Exclusion Criteria:

* Participant opposing or whose parents oppose participation of this children in the protocol.
* Patients under guardianship

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 participants, 500 children and 500 adults. All with at least one diagnosed specific learning disability
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Characterization of sleep disorders assessed using the Sleep Disturbances Scale for Children (SDSC) questionnaires in children | Baseline
  Scores are obtained after completing the different subsections of the questionnaire. The subsections represent the different sleep disorders. The scores obtained in the different subsections define whether a disorder is present or not.
Characterization of sleep disorders assessed using the Pittsburg Sleep Quality Index score in adults | Baseline
  Scores are obtained after completing the different subsections of the questionnaire. The subsections represent the different sleep disorders. The scores obtained in the different subsections define whether a disorder is present or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France